CLINICAL TRIAL: NCT03695757
Title: Evaluation of Immunostimulatory Effect of Intramuscular Administration of Autologous Total IgG in Human for Development of a New Immunotherapy
Brief Title: Development of a New Immunotherapy Using Intramuscular Administration of Autologous Total IgG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Dong-Ho Nahm, Professor, Ajou University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-THE-18-236
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Immunotherapy
Keywords: Immunoglobulin G; Treatment; Immunostimulatory effect; Tumor; Solid tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Intramuscularly administrations of autologous total IgG in healthy subjects and patients with advanced solid tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A) Healthy subjects (Experimental): Part A) Autologous total IgG 50mg will be administered to the healthy subjects by intramuscular injections, twice a week for 4 weeks (total 8 injections).
  Interventions: Biological: Part A) Healthy subjects
- Part B) Advanced solid tumor (Experimental): Part B) Autologous total IgG 50mg will be administered to the patients with advanced solid tumor by intramuscular injection, twice a week for 4 weeks (total 8 injections).
  Interventions: Biological: Part B) Advanced solid tumor

INTERVENTIONS:
Biological: Part A) Healthy subjects — Part A) Autologous total IgG 50mg will be administered to the healthy subjects by intramuscular injections, twice a week for 4 weeks (total 8 injections).
  Other Names: Intramuscular injections of autologous total IgG
  Arms: Part A) Healthy subjects
Biological: Part B) Advanced solid tumor — Part B) Autologous total IgG 50mg will be administered to the patients with advanced solid tumor by intramuscular injection, twice a week for 4 weeks (total 8 injections).
  Other Names: Intramuscular injections of autologous total IgG
  Arms: Part B) Advanced solid tumor

SUMMARY:
The purpose of this prospective pilot clinical study is to evaluate the safety and immunostimulatory effect of intramuscularly administrations of autologous total IgG (autologous total IgG therapy) in healthy subjects and patients with advanced solid tumor (non-small cell lung cancer, stomach cancer, colon cancer, ovarian cancer, breast cancer, pancreatic cancer, biliary cancer, melanoma, renal cell carcinoma etc.). In addition, antitumor effect of intramuscularly administrations of autologous total IgG in patients with advanced solid tumor will be also evaluated.

DETAILED DESCRIPTION:
After providing informed consent, study participants will be assessed for study eligibility at the screening visit. At screening visit (week -4), venous blood (320~400 mL) will be sampled using a double blood bag containing anticoagulant. Autologous plasma will be separated from the venous blood by centrifugation. During the 4 weeks of screening period, autologous total IgG (purity ≥97%) will be aseptically purified from the autologous plasma by chromatography using Protein A. Participants will receive the 8 intramuscular injections of autologous total IgG, twice a week for 4 weeks from baseline (week 0).

The investigators will evaluate the safety and immunostimulatory effect of intervention of this study by analyzing side effects, serum concentrations of immunological parameters (immunoglobulin, cytokine, etc.), and lymphocyte fraction by flow cytometry analysis of peripheral blood mononuclear cells.

[Part A) Autologous total IgG therapy in healthy subjects] The duration of this clinical study in healthy subjects is 16 weeks from the screening visit. A 4-week screening period will be followed by a 4-week intervention period and an 8-week follow-up period.

[Part B) Autologous total IgG therapy in patients with advanced solid tumor] The duration of this clinical study in patients with advanced solid tumor is 12 weeks from the screening visit. A 4-week screening period will be followed by a 4-week intervention period and a 4-week follow-up period(1 cycle).

If the patients agree to participate in additional long-term repeated study interventions at the end of 1st cycle of visit, patients will receive repeated study interventions in same the schedule up to week 44 (maximum 4 cycles). At the end of each cycle, antitumor effect will be evaluated by serum tumor marker concentrations, anatomical imaging, and Response Evaluation Criteria in solid tumors (RECIST ver. 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 19 years or older
2. Meeting the criteria for autologous blood donation 1) Body weight ≥32 kg (satisfying body weight limitation for planned sampling of 320 mL of venous blood volume) 2) Hemoglobin: ≥ 9 g/dL (Healthy volunteers Hemoglobin: ≥ 11 g/dL)
3. Provide signed informed consent
4. [Only for patients with advanced solid tumor] Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2 at the time of study enrollment.
5. [Only for patients with advanced solid tumor] Patients with a life expectancy longer than 3 months and metastatic (stage Ⅲ, Ⅳ) advanced solid tumor (non-small cell lung cancer, stomach cancer, colon cancer, ovarian cancer, breast cancer, pancreatic cancer, cholangiocarcinoma, malignant melanoma, renal cell carcinoma, etc.)
6. [Only for patients with advanced solid tumor] One or more target lesions must be present as confirmed by anatomical imaging (X-ray, CT sacn, MRI, etc.)

Exclusion Criteria:

1. Subjects under the age of 19 year, or unable to agree on their own (emergency patients, patients with mental disability, patients with limited capacity to consent due to stroke or delirium caused by diabetes), or severe disease whose expected survival duration is less than 3 months
2. Pregnancy or planned pregnancy within 1 year
3. Subjects who participated on another investigational device or drug studies within 4 weeks prior to screening visit
4. Medical history of alcohol or drug abuse within 2 years of the screening visit
5. Subjects is a member of the investigational team
6. Unable to comply with all clinic visits and study-related procedures
7. Planned or anticipated major surgical procedure within 4 weeks prior to baseline visit
8. [Only for patients with advanced solid tumor] A well-treated patients in combination with surgery and radiotherapy
9. [Only for patients with advanced solid tumor] Uncontrolled infections (bacterial, viral, fungal infection)
10. [Only for patients with advanced solid tumor] Has known active brain metastases(except for subjects with adequate treated and neurological asymptomatic at least 2 weeks, subjects without neurological symptoms without treatment for brain metastases, also subjects must be either off corticosteroid for corticosteroid therapy, or who have received stable doses of prednisone less than 10mg daily or who have received reduced doses may be enrolled.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with severe adverse events (AEs), serious adverse events (SAEs), treatment-related AEs, deaths, or discontinuation of study intervention due to AEs in healthy subjects | From baseline to week 12
Number of participants with severe adverse events (AEs), serious adverse events (SAEs), treatment-related AEs, deaths, or discontinuation of study intervention due to AEs in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year

SECONDARY OUTCOMES:
Number of participants with abnormal serum chemistry results and blood test results due to clinical study in healthy subjects | From baseline to week 12
Serum concentrations of immunological parameters (immunoglobulin, cytokine, etc.) in healthy subjects | From baseline to week 12
Lymphocyte fraction by flow cytometry analysis of peripheral blood mononuclear cells in healthy subjects | From baseline to week 12
Levels of cytokines secreted from peripheral blood cells in healthy subjects | From baseline to week 12
Quality of life (5-level EuroQoL Group's 5-dimension; EQ-5D-5L) in healthy subjects | From baseline to week 12
  The 5-level EuroQoL Group's 5-dimension (EQ-5D-5L) consists of 2 parts: the descriptive system and the EQ visual analogue scale (VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of perceived problems: no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems. In addition, the EQ-5D-5L include an EQ-VAS where the endpoints are labeled on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Subjective index of pain and fatigue (Visual Analogue Scale; VAS, Numeral Rating Scale; NRS) in healthy subjects | From baseline to week 12
  The 100-mm Visual Analogue Scale (VAS) ranges from 0 (absent) to 10 (worst imaginable). The 11-point Numerical Rating Scale (NRS) ranges from 0 (absent) to 10 (worst imaginable).
Number of participants with abnormal serum chemistry results and blood test results due to clinical study in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Serum concentrations of immunological parameters (immunoglobulin, cytokine, etc.) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Lymphocyte fraction by flow cytometry analysis of peripheral blood mononuclear cells in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Levels of cytokines secreted from peripheral blood cells in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Objective response rate (ORR) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Disease control rate (DCR) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Duration of response (DOR) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Progression-free survival (PFS) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Overall survival (OS) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
The tumor marker concentrations in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
Quality of life (5-level EuroQoL Group's 5-dimension; EQ-5D-5L) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
  The 5-level EuroQoL Group's 5-dimension (EQ-5D-5L) consists of 2 parts: the descriptive system and the EQ visual analogue scale (VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of perceived problems: no problems, slight problems, moderate problems, severe problems, and unable to/extreme problems. In addition, the EQ-5D-5L include an EQ-VAS where the endpoints are labeled on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Subjective index of pain and fatigue (Visual Analogue Scale; VAS, Numeral Rating Scale; NRS) in patients with advanced solid tumor | From baseline to week 8 and through study completion, an average of 3 year
  The 100-mm Visual Analogue Scale (VAS) ranges from 0 (absent) to 10 (worst imaginable). The 11-point Numerical Rating Scale (NRS) ranges from 0 (absent) to 10 (worst imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ho Nahm, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university hosiptal, Suwon, Gyeong-gi Do, South Korea

REFERENCES:
- [Derived] Kwon B, Yang SJ, Cho SM, Kim ME, Nahm DH. Intramuscular administration of autologous total immunoglobulin G induces immunomodulatory effects on T cells in healthy human subjects: An open-labeled prospective single-arm trial. Medicine (Baltimore). 2022 Jun 3;101(22):e29486. doi: 10.1097/MD.0000000000029486. PMID 35665739